CLINICAL TRIAL: NCT05527483
Title: Digital PET/CT Using [Ga-68]PSMA vs. [F-18]NaF for Evaluation of Osseous Metastatic Involvement in Prostate Cancer Patients
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Norbert Avril, Division Chief, Nuclear Medicine, University Hospitals Cleveland Medical Center
Other Study IDs: STUDY20220121
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer
Keywords: Bone Metastasis; PET/CT
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11; Sodium Fluoride; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- [F-18]NaF: Patients will receive 8-12 mCi of [F-18]NaF delivered as an intravenous (IV) bolus injection, followed by digital PET/CT imaging.
  Interventions: Drug: [68Ga]PSMA; Drug: Flourine-18 [F-18] Sodium Fluoride (NaF); Diagnostic Test: PET/CT
- [Ga-68]PSMA: Patients will receive up to 6 mCi of [Ga-68]PSMA delivered as an intravenous (IV) bolus injection, followed by digital PET/CT imaging
  Interventions: Drug: [68Ga]PSMA; Drug: Flourine-18 [F-18] Sodium Fluoride (NaF); Diagnostic Test: PET/CT

INTERVENTIONS:
Drug: [68Ga]PSMA — Patients will receive up to 6 mCi of [Ga-68]PSMA delivered as an intravenous (IV) bolus injection, followed by digital PET/CT imaging
Drug: Flourine-18 [F-18] Sodium Fluoride (NaF) — Patients will receive 8-12 mCi of [F-18]NaF delivered as an intravenous (IV) bolus injection, followed by digital PET/CT imaging.
Diagnostic Test: PET/CT — Patients will receive [68Ga]PSMA with a PET/CT and Flourine-18 [F-18] Sodium Fluoride (NaF) with a PET/CT

SUMMARY:
The purpose of this study is to evaluate a radioactive diagnostic study drug, which is called Gallium-68 Prostate Specific Membrane Antigen ([Ga-68]PSMA) for detection of bone metastasis in patients with prostate cancer.

For imaging the investigators will use a FDA approved imaging technology, digital Positron Emission Tomography (PET/CT). The investigators would like to know if digital PET/CT using [Ga-68]PSMA provides accurate information about the extent of bone metastases.

Therefore, the investigators will compare[Ga-68]PSMA PET/CT with Flourine-18 [F-18] Sodium Fluoride (NaF), which is a high resolution bone scan. [F-18]NaF is FDA approved and the reference standard for evaluating the presence of bone metastases.[Ga-68]PSMA is an investigational (experimental) drug that works by binding to Prostate Specific Membrane Antigen, which is overexpressed in prostate cancer. [Ga-68]PSMA is experimental because it is not approved by the Food and Drug Administration (FDA) at University Hospitals. However, FDA approval has been obtained for this study protocol by an Investigational New Drug (IND) application.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients must have a history of prostate cancer
* 2) Patients have known or highly suspected osseous metastatic involvement defined by the referring physician based on clinical history and/or findings from standard of care imaging.
* 3) Patients ≥ 18 years old
* 4) Patients able to tolerate PET/CT scans
* 5) Informed written consent must be given and signed

Exclusion Criteria:

* 1. Subjects who do not meet the noted inclusion criteria
* 2. Patients < 18 years old
* 3. Subjects who refuse to give or are unable to sign the informed consent
* 4. Anti-cancer treatment (chemotherapy and/or radiation therapy) within the last 2 weeks
* 5. Patients with a known allergy against Ga-68 PSMA or F-18 NaF

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Study Population: Members of all races and ethnic groups are eligible for this trial. Due to the nature of the disease, only people being diagnosed with prostate cancer are eligible.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Uptake of [Ga-68]PSMA as measured by lesion by lesion analysis | Up to 90 minutes
  Classified using a 5-point score with one being definitely metastatic and five being definitely benign

SECONDARY OUTCOMES:
Focally increased [Ga-68]PSMA uptake as measured by PET/CT | Up to 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jones, M.D., Principal Investigator — UH, Cleveland Medical Center; Norbert Avril, M.D., Principal Investigator — UH, Cleveland Medical Center
Locations (1):
- Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No